CLINICAL TRIAL: NCT00065416
Title: Evaluating Therapeutic Massage for Chronic Neck Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: R21AT001584-01 (NIH)
Record Dates: First submitted 2003-07-22; First posted 2003-07-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-10

CONDITIONS: Neck Pain; Cervicalgia
Keywords: neck pain; cervicalgia; massage
MeSH Terms: conditions — Neck Pain | interventions — Massage

INTERVENTIONS:
Procedure: massage

SUMMARY:
This study will provide the basis for a full-scale trial to evaluate the effectiveness and safety of therapeutic massage for chronic neck pain (CNP).

DETAILED DESCRIPTION:
Neck pain is one of the most common problems affecting the health of Americans and is a leading reason for using complementary or alternative medical (CAM) therapies. Therapeutic massage is one of the most popular CAM treatments for neck pain, but little is known about its effectiveness. This study will lay the groundwork for a full-scale trial that evaluates the effectiveness of therapeutic massage for chronic neck pain.

The study will involve two phases. During Phase I, researchers will develop and pre-test key components for a randomized clinical trial. In Phase II, the safety and efficacy of massage for CNP will be evaluated. The changes in symptoms, function, and quality of life in massage and self care groups will be evaluated midway through treatment, at the end of treatment and at 6 months post randomization.

ELIGIBILITY:
The inclusion and exclusion criteria will be developed through consultation with a medical expert on neck pain and several massage consultants

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Sherman, PhD, Principal Investigator — Group Health Cooperative Center for Health Studies
Locations (1):
- Group Health Cooperative, Center for Health Studies, Seattle, Washington, United States